CLINICAL TRIAL: NCT06173128
Title: Alteration of Respiratory Microbiota and Local Immune Response in Common Variable Immunodeficiency
Brief Title: Respiratory Microbiota and Immune Response in CVID
Status: Recruiting | Type: Observational
Sponsor: Boston University (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: H-42779
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: CVID
Keywords: Impaired antibody response; Pattern recognition receptor; Immunoglobulins; Respiratory microbiota; Nuclear Factor Kappa B (NF-κB)-driven cytokines; Complex microbial-host cell interactions; Pulmonary biology; RNAseq analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, saliva, nasopharyngeal, and sputum samples will be collected. 50 ml of blood will be collected/participant.This collection of blood will constitute the study biological sample repository. Peripheral blood mononuclear cells (PBMCs) plasma samples will be used for flow cytometry, cell culture, and enzyme-linked immunosorbent assays. RNAseq will be done on nasopharyngeal samples. Sputum samples will have measurement of lymphocyte subsets (by flow cytometry), cytokines and immunoglobulins (by multiplex ELISA), and RNA (both bacterial and host by RNA sequencing) in the laboratory.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Antibody deficient participants: Provider referred patients that have antibody deficiency.
- Controls: Patients without antibody deficiency from the allergy and immunology clinic at Boston Medical Center and from healthy volunteers at the BU School of Medicine.

SUMMARY:
Common variable immunodeficiency (CVID) is the most prevalent symptomatic primary immunodeficiency. Respiratory ailments are the most frequent complications of CVID, with chronic pulmonary disease developing in 30-60% and even more experiencing frequent acute respiratory infections. This project aims to establish cutting-edge approaches to study pulmonary biology in CVID and apply novel bioinformatics strategies to study complex interactions among microbes and host cells by direct sampling of the respiratory tract. The central hypothesis for this research is that antibody (Ab) deficiency in CVID alters respiratory microbiota and host interactions to drive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary antibody deficiency diagnosed by their treating physician
* Controls will not have a diagnosis of immunodeficiency of any sort
* Male and female patients will be enrolled evenly

Exclusion Criteria:

* Patients who self identify as pregnant
* Patients with asthma or chronic obstructive pulmonary disease (COPD) that are not well controlled clinically

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be enrolled from the Boston Medical Center allergy and immunology clinics and from healthy volunteers at the Boston University medical campus (BUMC). They will be assigned into one of two groups: antibody deficient patients and controls. Blood, nasopharyngeal swab, saliva, and sputum (if possible) samples will be collected from each participant, ideally on the same day.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Feasibility of respiratory sample RNA sequencing (RNAseq) analysis | 1 year
  Quality control analysis of RNA samples collected from nasopharyngeal swabs for adequacy to perform RNA-seq analysis will be performed. This will be done using the Boston University (BU) Medical Campus RNA core facility bioanalyzer, which will assess for adequate RNA quality and quantity for RNA-seq
Analysis of saliva sampling | 2 years
  Saliva samples will be analyzed by enzyme-linked immunosorbent assay (ELISA) and multiplex analysis (Luminex) for levels of antibodies as well as cytokines and other inflammatory proteins.
Respiratory microbiota analysis by RNA-seq of nasopharyngeal samples | 2 years
  RNA-seq data derived from nasopharyngeal samples will undergo computational analysis to identify alterations of microbiota constituency.
Host gene expression analysis by RNA-seq of nasopharyngeal samples | 2 years
  RNA-seq data derived from nasopharyngeal samples will undergo computational analysis to identify alterations of host gene and pathway expression.

SECONDARY OUTCOMES:
Altered respiratory microbiota due to primary antibody deficiency | 2 years
  RNA seq will be used to determine if primary antibody deficiency alters respiratory microbiota
Altered gene expression due to primary antibody deficiency | 2 years
  RNA seq will be used to determine if primary antibody deficiency alters host gene expression.

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Maglione, MD PhD, Principal Investigator — Boston University Chobanian & Avedisian School of Medicine, Pulmonary Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided